CLINICAL TRIAL: NCT05912478
Title: The Effect of Video-Based Game Therapy on Activation of Scapular Muscles in Children with Thoracic Hyperkyphosis
Brief Title: Video-Based Game Therapy in Thoracic Hyperkyphosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Assos. Prof, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001-PhD
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-07

CONDITIONS: Hyperkyphosis; Postural Kyphosis; Exergaming; Muscle Weakness; Muscle Tightness; Posture Disorders in Children
Keywords: video games; hyperkyphosis; stability; sapula; muscle activation; posture
MeSH Terms: conditions — Kyphosis; Muscle Weakness | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Videogame-Based Therapy Games for the Nintendo Switch (Version 2) will be used for eight weeks, three days per week, for a total of 24 sessions.
  Interventions: Other: Videogame-Based Therapy
- Control Group (Other): The participants on the waiting list will be evaluated as the control group. For eight weeks, the control group will be instructed to maintain their daily routine.
  Interventions: Other: Waiting list

INTERVENTIONS:
Other: Videogame-Based Therapy — The Nintendo Switch (Version 2) will be used to play video games. Within the scope of the study, Nintendo Switch games were analyzed with respect to their technical and fictional characteristics, required and optional movement patterns, difficulty levels, transitions between difficulty levels, and compatibility with priority problems. The selected activities will prioritize the activation of the scapular muscles. Throughout the activities, the participant will be required to mimic the on-screen avatar's movements. The player will receive a higher score if his or her movements in the game resemble the avatar's in terms of angular, velocity, and fluidity.
  Arms: Study group
Other: Waiting list — The participants who were placed on a waiting list for eight weeks and constituted the control group will be asked to carry on with their normal activities. Participants in the control group will be contacted by phone in the fourth week to inquire about their status and to remind them that the exercise program will begin in the coming weeks. At the end of the 8-week study, the participants from the control group will participate in the exercise program.
  Arms: Control Group

SUMMARY:
The scapula provides the base of the kinetic chain, which is stabilized by the surrounding muscles. Considering that activating the scapular musculature to stabilize the spine would restore the relationship between body segments, analyzing the scapular muscle activations in the treatment of hyperkyphosis may be a crucial component of an effective therapeutic program.

Video games can be used to stimulate scapular muscles in children with thoracic hyperkyphosis because a game-based exercise program has been observed to increase voluntary motor control in children, thereby promoting selective muscle activation. The purpose of this study is to investigate the impact of video game therapy on the activation of scapular muscles and postural stability in children with thoracic hyperkyphosis, as well as the contribution of these variables to upper extremity performance.

DETAILED DESCRIPTION:
Postural hyperkyphosis is a common spine curvature that develops when individuals with inadequate overall muscular strength are continuously exposed to high-intensity external stresses while standing. It is a deformity frequently observed in healthy children and adolescents, but it is often overlooked and can be detected through school examinations. Postural hyperkyphosis has significant effects on a person's overall health, physical performance, and quality of life. When the angle of kyphosis increases, it causes severe health problems, such as sensitivity in the spine, tension, neck, waist, and back discomfort. Untreated hyperkyphosis, which begins in childhood and persists into adulthood, has the potential to increase healthcare costs. It is crucial to control this deformity during childhood and adolescence, given the increase in the incidence of hyperkyphosis due to an increasing reliance on technology and its negative health and economic consequences. In addition to angular correction of the deformity, the entire spine within the kinetic chain should be examined when treating postural hyperkyphosis.

In clinical practice, it is common to convey exercise routines to children as enjoyable activities. In accordance with technological advancements, game-based exercise regimens are now also available as software. In conventional physiotherapy programs, the motivation, willingness to persist, and active participation of children gradually decline. Making it more challenging for the physiotherapist to motivate children to exercise and assure the program's sustainability. Nonetheless, it is vital to maintain enthusiasm throughout this lengthy treatment process, particularly in chronic conditions such as hyperkyphosis.

On the basis of the inclusion and exclusion criteria, individuals diagnosed with thoracic hyperkyphosis who required rehabilitation but did not receive spinal region treatment will be recruited to participate in the study. Random assignment will designate participants to either the study group (video-based game therapy) or the control group (waiting list).

The demographic and clinical characteristics of both groups will be evaluated, along with muscle activation, muscle strength, muscle tone, rigidity, posture, perception of cosmetic deformity, upper extremity performance, physical activity levels, treatment satisfaction, and exercise adherence. The study group volunteers will be required to participate in 24 sessions, three times per week for eight weeks, comprising of games selected at the conclusion of the initial evaluation session. The Nintendo Switch will be used for playing video games. After the initial evaluation, all subjects in the control group will be placed on an eight-week waiting list. At the end of the study, the control group participants will engage in the same exercise regimen.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic kyphosis angle (Cobb): ≥40˚- <65˚ on lateral radiograph
* Age between 7-18 years

Exclusion Criteria:

* Those with congenital or rigid deformity/anomaly in the spinal area
* Those who have had major surgery or trauma related to the musculoskeletal system, especially the spinal region
* Those who received physiotherapeutic intervention in the spinal region in the last 6 months
* Those who use corsets
* Having a BMI ≥30
* Those who are interested in sports in which the upper extremity is regularly used actively (swimming, volleyball, tennis, handball, etc.) Those who have visual problems and are sensitive to light.
* Those with vestibular problems (Unterberger test positive)
* Those with hearing problems
* Those who have difficulty perceiving the given commands
* Those with systemic diseases (Diabetes, hypothyroidism, infection, malignancy...)
* Those with neurological disease
* Those with rheumatic disease in the active phase

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Muscle Activation | 8 weeks
  The electrical activity of the muscle during rest and contraction is called electromyogram, and recording this activity is called electromyography (EMG). Superficial EMG (yEMG) is preferred in physiotherapy and rehabilitation researches due to its noninvasive nature, no risk of infection and ease of use. In our study, Noraxon Myosystem (Noraxon Inc., Scottsdale, AZ, USA) yEMG will be used to measure the electrical activity of the upper, middle and lower trapezius, pectoralis major, and serratus anterior muscles. Electrodes will be placed in orientation parallel to the identified muscle fibers as recommended by "Surface ElectroMyoGraphy for the Non-Invasive Assessments of Muscles SENIAM)". Activations of these muscles will be recorded as a percentage of maximum voluntary isometric contraction (%MVIC). In addition, analyzes will be made about fatigue, coactivation and activation time of the muscles.
Muscle Tone and Stiffness | 8 weeks
  MyotonPRO (Muomeetria Ltd., Tallinn, Estonia) will be used to measure the tone and stiffness of the upper, middle and lower trapezius, pectoralis major and serratus anterior muscles. Myotonometry reflects the viscoelastic properties of the muscle such as tone and stiffness by creating oscillation in the muscle fiber and is an acceptable and reliable method for measuring the mechanical properties of the muscles. In our study, after the participants rest for 5 minutes, the arms will be left relaxed in the sitting position and the measurement will be taken from the most swollen part of the relevant muscles. During the measurement, the test probe of the myotonometer will be placed vertically on the skin surface. The measurement will be started by pushing the probe to the required depth on the skin surface. Whether the required depth has been reached or not will be checked by turning the indicator light on the device from red to green.
Posture | 8 weeks
  PostureScreen Mobile software is a valid and reliable application that evaluates the changes in a person's posture. In our study, the evaluation of frontal and sagittal plane posture will be calculated by marking reference points on the photographs taken from the front, back and sides of the patient in the PostureScreen Mobile application.Photographing, positioning and determination of reference points of the participants will be standardized. During the photo shoot, the feet of the participants will be positioned bare and parallel to each other, attention will be paid to the absence of clothing and the bulk of the hair so that the reference points are clear. During the shoot, participants will be asked to keep their arms loose and look straight ahead.
Satisfaction with Body Image | 8 weeks
  Since there is no scale specific to hyperkyphosis deformity in the literature that evaluates individuals' own perception of cosmetic deformity, a numerical rating scale with values between 0-10 will be used to evaluate how the perception of cosmetic deformity changes.
Perception of Spinal Deformity | 8 weeks
  Perception of spinal deformity will be assessed with the Kyphosis-Specific Spinal Appearance Questionnaire.The Kyphosis Specific Spinal Appearance Questionnaire has been developed to assess appearance in hyperkyphosis patients. The KSAQ included 10 items on a Likert scale (1 to 5) regarding patients' perceptions of appearance, with higher scores indicating worsening deformity and greater kyphosis-specific appearance concern
Medicine Ball Throwing Test | 8 weeks
  It will be used to evaluate the explosive power of the upper extremity. Participants will be positioned in a chair without armrests in an upright position with their ankle, knee and hip joints at 90 degrees. He will be asked to grasp the 3 kg medicine ball with both hands and throw it forward over the head without bending his body forward and without flexing his elbows. The first point where the ball touches the ground will be measured from the starting point and the value will be recorded in cm. The test will be repeated three times and the average of the values recorded. The test of the participants will be invalidated and the test will be repeated if they throw the ball down to the level of their neck or make the throw by leaning forward from the trunk.
Closed Kinetic Chain Upper Extremity Stability Test | 4 months
  It will be used to evaluate upper extremity strength, endurance and closed kinetic chain. The test will also be performed following the guidelines described by Oliveira et al. During the test, male participants will be placed in the push-up position, and female participants in the modified push-up position (with knee support), on 2 tapes glued to the floor with a distance of 90 cm between the two hands. Participants will be asked to touch the other hand with one hand while maintaining the push-up position for 15 seconds, and the number of reps completed for the right and left will be recorded. The test will be repeated three times and the average of the values recorded. There will be 45-second rest breaks between each test. In the test-retest reliability study of the test in adolescents, the intraclass correlation coefficient (ICC) was found to be 0.68.
Scapular Endurance Test | 8 weeks
  The endurance of the scapular muscles will be evaluated with the Scapular Muscular Endurance Test. The Scapular Muscular Endurance Test will be performed with the participants facing the wall in a standing position, with the shoulders and elbows in the 90° flexion position. With both scapulae in neutral position, the participant will place the most appropriate length of 10 wooden sticks (18-36 cm) between their elbows and a dynamometer between their hands. While in this position, the participant will be asked to perform external rotation of the shoulder and maintain this force until a load of one kilogram is reached on the dynamometer, and the results will be recorded in seconds. The test will be terminated if the participant is unable to maintain the applied resistance, drops the bar between their elbows, or is unable to maintain 90 degrees of shoulder flexion and becomes unbearable
Reaction time | 8 weeks
  Nelson Hand Reaction Test will be used to evaluate reaction speed. The test is performed while the subject sits in a chair, placing his hands on the table's edge with the palms facing each other. The little fingers of both hands are in contact with the edge of the table and there is a distance of 30 cm between them. The therapist holds the wooden ruler at the midpoint of the subject's fingers. The ruler is left after the subject gains attention with the therapist's "Ready" command (0.5-2 seconds). The subject holds the ruler by squeezing it between both hands with a horizontal movement as soon as possible. Once the ruler is captured, the reading at the point just above the top edge of the hand is recorded.

SECONDARY OUTCOMES:
Demographic and Clinical Characteristics | 8 weeks
  Demographic and clinical characteristics of the participants will be recorded with an evaluation form consisting of 2 parts. In the first part, demographic information such as age, gender, height, weight, waist circumference, dominant side, whether there is a sport branch of interest will be questioned. In the second part, clinical features such as radiography (Cobb angle), spine alignment (flexicurve ruler and wall-occiput distance), pain (Numeric Grading Scale) will be recorded.
Flexicurve Rule | 8 weeks
  Flexicurve Ruler is a non-invasive, plastic, easily shaped and easily accessible, valid and reliable tool used to get an idea about the curvature of kyphosis. In our study, C7 and T12 reference points will be accepted as the starting and ending points, and pressure will be applied towards the caudal so that the flexible ruler takes the shape of the curvature. The width and height measurements of the formed shape will be recorded in cm.
Wall-Occiput Distance Measurement: | 8 weeks
  For Wall-Occiput Distance measurement, participants will be asked to touch their occiput to the wall with their back and heels against the wall and head forward. The presence of hyperkyphosis will be considered positive if the wall cannot be touched with the occiput. During the measurement, two rulers will be used. The first ruler will be placed on the occiput parallel to the ground, and the second ruler will be placed between the first ruler and the wall to measure the perpendicular distance. The measurement will be repeated three times in succession with a short rest period, and the average values will be recorded.
The Numerical Rating Scale | 8 weeks
  The Numerical Rating Scale is a simple, sensitive and reproducible tool that is often used to assess pain severity. It has become the most frequently used self-assessment scale in studies due to its easy application. On this scale, patients will be asked to rate the severity of their pain between 0 and 10, with 0 being "no pain" and 10 "unbearable pain". In the first evaluation and the second evaluation after the treatment, all participants will be questioned about rest, activity and night pain in the last 6 months.
Muscle Strength | 8 weeks
  In our study, maximal isometric muscle strength will be measured with a hand-held dynamometer (Lafeyette Instrument, Lafayette, IN), which has been shown to be valid and reliable. In our study, participants will be placed in standardized positions and maximal voluntary isometric muscle strength will be measured for bilateral trapezius upper-middle-lower fibers, levator scapula, pectoralis major, rhomboid and serratus anterior muscles. For each muscle, 3' measurements would be made and their average values (kg/N) would be recorded.
Physical Activity Level | 8 weeks
  The physical activity level of the cases will be evaluated with the Child Physical Activity Questionnaire, which is frequently used in the clinic and whose validity and reliability studies have been conducted. This questionnaire is a 5-point Likert-type questionnaire consisting of 9 items in total, questioning the physical activities done in the last 7 days and the frequency of these activities. A high score indicates an increased level of physical activity.
Treatment Satisfaction | 8 weeks
  The level of satisfaction with the treatment received by all participants at the end of the study will be evaluated with the "Global Rating of Change Scale". The Global Rating of Change Scale is a scale by which patients determine the amount of improvement or worsening in their health status over time from their own perspective. There are different types of ratings in Global Rating of Change Scale. In our study, the form consisting of 7 levels in the -3 and +3 value ranges (-3: I am much worse, 0: I am the same, +3: I am completely cured) will be preferred.
Exercise Adaptation | 8 weeks
  In order to evaluate the exercise compliance of the participants participating in the study, the number of days they participated in video-based game therapy during 8 weeks, the screen time they spent playing games in each session, the number of listening sessions and times they gave in one session and between games will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zengin Alpozgen, Asst. Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No